CLINICAL TRIAL: NCT03153384
Title: Impact of the Blood Culture Technique on the Diagnosis of Infectious Diseases: Case of Infective Endocarditis.
Brief Title: Impact of the Blood Culture Technique on the Diagnosis of Infective Endocarditis
Acronym: UniEndo
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GOEHRINGER François, Dr, Central Hospital, Nancy, France
Other Study IDs: APJ2015/UNIENDO-GOEHRINGER/SKJ
Record Dates: First submitted 2017-05-05; First posted 2017-05-15 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Bacteremia; Infective Endocarditis
Keywords: Diagnosis; Blood Culture
MeSH Terms: conditions — Bacteremia; Endocarditis; Disease | interventions — Blood Culture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one both experimental and control arm: Each patient experiences two methods of blood cultures.
  Interventions: Procedure: Blood Culture

INTERVENTIONS:
Procedure: Blood Culture — For each patient, one single high volume blood culture (3 aerobic and 3 anaerobic of 8 to 10 mL each, numbered), and then 2 samples of 16 to 20 mL (one aerobic bottle and one anaerobic for each sample).

SUMMARY:
To evaluate the performance of a single high volume blood culture sampling strategy versus the actually used multiple sampling strategy for the diagnosis and categorization of infective endocarditis according to the Duke-Li classification in a Population of adults suspected of infective endocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Suspected endocarditis: Patients with Duke-Li-ESC 2015 classification as a major morphological criterion or at least two minor criteria, other than a microbiological criterion, will be considered suspicious of infectious endocarditis.
* Not objecting to their inclusion in the study after delivery and explanation of the information form.
* Absence of microbiological documentation sought or available at the time of inclusion (a patient having already had negative blood cultures or being identified during the screening can be included).

Exclusion Criteria:

* Antibiotherapy adapted to a situation of endocarditis, introduced more than 24 hours or stopped for less than 7 days in case of therapeutic window.
* Any previous antibiotic therapy in the 7 days preceding the inclusion leading to an improvement in the clinical symptomatology.
* State of consciousness not allowing loyal information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult patients suspected of infective endocarditis
Sampling Method: Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Compared performance of a single high volume blood culture vs. multiple blood culture of usual volume for the diagnosis of infective endocarditis | At the end of the hospitalization, or at the time of death if occurred during hospitalization; i.e. an average of 6 weeks after the inclusion
  Sensitivity/Specificity/Accuracy of positive bloodculture sets vs. final diagnosis assessed by the medical team (gold standard)

SECONDARY OUTCOMES:
Diagnostic performance of the single high volume blood culture for the diagnosis of infective endocarditis | At the end of the hospitalization, or at the time of death if occurred during hospitalization; i.e. an average of 6 weeks after the inclusion
  according to the level of suspicion of infective endocarditis, the type of microorganism involved, the underlying cardiopathy.
Measuring the nursing time required for both sampling methods. | At T0, i.e. at the inclusion of the patient
  Time for blood culture setting, processing and sending
Diagnosis of infective endocarditis: confirmed, possible or excluded | At the end of the hospitalization, or at the time of death if occurred during hospitalization; i.e. an average of 6 weeks after the inclusion
  Applying the Classification of Duke-Li according to the modified diagnostic criteria of the European Society of Cardiology Recommendations 2015.

CONTACTS AND LOCATIONS:
Overall Officials: François Goehringer, MD, Principal Investigator — Centre Hospitalier Universitaire de Nancy, Nancy, France; Xavier Duval, MD PhD, Study Chair — APHP, Hôpital Bichat Claude Bernard, Paris, France.; Christine Selton-Suty, MD, Study Chair — Centre Hospitalier Universitaire de Nancy, Nancy, France; Nejla Aissa, MD, Study Chair — Centre Hospitalier Universitaire de Nancy, Nancy, France
Locations (8):
- France (8):
  - Hôpital Nord Franche Comté, Belfort
  - Centre Hospitalier universitaire de Besançon, Besançon
  - Centre Hospitalier universitaire de Dijon, Dijon
  - Centre hospitalier Universitaire de Nancy, Nancy
  - Hopital BIchat Claude Bernard, Paris
  - Centre Hospitalier Universitaire de Reims, Reims
  - Centre Hospitalier Univesitaire de Rennes, Rennes
  - Hôpitaux Civils de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arendrup M, Jensen IP, Justesen T. Diagnosing bacteremia at a Danish hospital using one early large blood volume for culture. Scand J Infect Dis. 1996;28(6):609-14. doi: 10.3109/00365549609037969. PMID 9060065
- [Background] Dargere S, Parienti JJ, Roupie E, Gancel PE, Wiel E, Smaiti N, Loiez C, Joly LM, Lemee L, Pestel-Caron M, du Cheyron D, Verdon R, Leclercq R, Cattoir V; UBC study group. Unique blood culture for diagnosis of bloodstream infections in emergency departments: a prospective multicentre study. Clin Microbiol Infect. 2014 Nov;20(11):O920-7. doi: 10.1111/1469-0691.12656. Epub 2014 Jun 14. PMID 24766148
- [Background] The 2015 ESC Guidelines for the management of infective endocarditis. Eur Heart J. 2015 Nov 21;36(44):3036-7. doi: 10.1093/eurheartj/ehv488. PMID 26590409
- [Background] Li JS, Sexton DJ, Mick N, Nettles R, Fowler VG Jr, Ryan T, Bashore T, Corey GR. Proposed modifications to the Duke criteria for the diagnosis of infective endocarditis. Clin Infect Dis. 2000 Apr;30(4):633-8. doi: 10.1086/313753. Epub 2000 Apr 3. PMID 10770721